CLINICAL TRIAL: NCT03498248
Title: Efficacy of Granulocyte-Colony Stimulating Factor (G-CSF) Related Clinical Implications in Cytotoxic Chemotherapy Induced Neutropenia
Brief Title: Efficacy of Granulocyte-Colony Stimulating Factor (G-CSF)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: DERSHENG SUN (Other)
Responsible Party: Sponsor-Investigator, DERSHENG SUN, Clinical Associated Professor, The Catholic University of Korea
Organization: The Catholic University of Korea (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Granulocyte-Colony Stimulating
Record Dates: First submitted 2018-04-07; First posted 2018-04-13 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Neutropenia
MeSH Terms: conditions — Neutropenia | interventions — Lenograstim

STUDY DESIGN:
Intervention Model Description: neutropenia after cytotoxic chemotherapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neutropenia in chemotherapy (Experimental): Neutropenia after cytotoxic chemotherapy
  Interventions: Drug: lenograstim

INTERVENTIONS:
Drug: lenograstim — injection of lenograstim in patients with neutropenia after cytotoxic chemotherapy

SUMMARY:
The purpose of this study was to analyze the clinical factors associated with the effect of Granulocyte-Colony Stimulating Factor (G-CSF).

DETAILED DESCRIPTION:
1. Granulocyte-Colony Stimulating Factor (G-CSF) G-CSF is known to be a synthetic cytokine that induces neutrophil differentiation and proliferation survival during leukocyte differentiation, and increases the activity in the periphery of mature neutrophils, which play an important role in human immunity. Cytotoxic chemotherapy inhibits bone marrow hematopoiesis. Inhibition of bone marrow hematopoiesis causes anemia, thrombocytopenia and leukopenia, and significant leukocytopenia causes opportunistic infection. G-CSF is an indispensable drug for the treatment of leukopenia caused by cytotoxic chemotherapy in solid and blood cancer patients receiving chemotherapy.
2. Chemotherapy with chemotherapy and G-CSF The severity of neutropenia induced by chemotherapy was grade 1 (<1500 / mm3), grade 2 (<1500-1000 / mm3) and grade 3 (<1000) based on the Common Terminology Criteria for Adverse Events To 500 / mm3) and grade 4 (<500 / mm3). Cytotoxic anticancer drugs used in general chemotherapy cause neutropenia, and febrile neutropenia occurs in 10-20% of patients. In order to recover this, grade 4 neutropenia with an absolute neutrophil count (ANC) of less than 500 and neutrophil to grade 2 or higher with G-CSF in case of febrile grade 3 neutropenia.
3. G-CSF dose and timing G-CSF (Renoglass team lenograstim 250 ug) was subcutaneously injected to a solid tumor (grade 3 or higher regardless of fever) with grade 3 or grade 4 neutropenia with fever Until then, take medication daily. It is used regardless of gender, age, weight, body mass index, method of using anticancer, and injection time.

However, the actual timing and extent of neutrophil recovery after G-CSF administration varies from patient to patient. G-CSF is a cytokine that is currently used in clinical trials. However, there are insufficient studies to investigate the clinical factors involved in the recovery of neutrophils in bone marrow after G-CSF administration in domestic cancer patients. Therefore, this study aims to analyze the clinical factors for the recovery of bone marrow hematopoietic function of G-CSF administered in neutropenia following cytotoxic chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with solid cancer and blood cancer
2. Patients who received chemotherapy with moderate risk (Appendix 1, Appendix 2)
3. CTCAE version 4.0 showed grade 4 neutropenia, grade 3 neutropenia (blood cancer), Decreased grade 3 neutrophils with fever (solid cancer)
4. Those who understand and agree with the purpose of the research

Exclusion Criteria:

* 1) Patients with hypersensitivity to G-CSF 2) Patients not diagnosed with hematologic tumor 3) grade 1, grade 2 or more neutropenia 4) Patients who did not sign a consent agreement

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2018-02-19 (Actual); Primary Completion 2018-08-31 (Estimated); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
duration of severe neutropenia | at least in 1 wk
  count days of neutrophils increased above 1,000

CONTACTS AND LOCATIONS:
Overall Officials: Yoon Ho Ko, Principal Investigator — Uijeongbu St. Mary's Hospital
Locations (1):
- the Catholic university of Korea, Seoul, Gyounggido, South Korea